CLINICAL TRIAL: NCT04356989
Title: Xarelto® for the Prevention of Stroke and Noncentral Nervous Systemic Embolism in Non-valvular Atrial Fibrillation With REnal Impairment in Taiwanese Population.
Brief Title: Study to Gain Information on the Drug Xarelto for the Prevention of Brain Attack and Blockage of an Artery in the Non-central Nervous System Due to Irregular Heartbeat in Taiwanese Patients Suffering From Decreased Renal Function
Acronym: XARETO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20901
Record Dates: First submitted 2020-04-21; First posted 2020-04-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Stroke
MeSH Terms: conditions — Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivaroxaban: Adult NVAF patients with renal impairment, who are prescribed with rivaroxaban to prevent stroke or non-central nervous system (CNS) systemic embolism (SE).
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — The adminstration dose is decided by the attending physician in advance based on the patients' CrCl and in compliance with local market authorization of rivaroxaban.

SUMMARY:
In this study researchers want to learn more about on the safety of the drug Xarelto. The study will enroll patients for whom the treating doctor are prescribing Xarelto for the prevention of brain attack or the prevention of blockage of an artery in the non-central nervous system. Only patients suffering from decreased renal function and irregular heart beat will be considered. The study plans to include 500 Taiwanese adult male and female patients with the age above 20 years. Patients will be followed up based on routine medical practice over a period of 12 months and information on their well-being and any medical events will collected.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 20 years of age
* Diagnosis of non-valvular atrial fibrillation (NVAF)
* Patients for whom the decision to initiate treatment with rivaroxaban is made as per physician's routine treatment practice
* Previously documented CrCl of 15-50 mL/min within 6 months before enrollment (last available value)

Exclusion Criteria:

* Contraindications for rivaroxaban according to the local market authorization/ Summary of Product Characteristics
* Patients participating in an investigational program with interventions outside of routine clinical practice.
* Planned treatment with other anticoagulants
* Expected renal-replacement therapy within the next 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of Taiwanese NVAF patients with documented CrCl of 15-50 mL/min, requiring rivaroxaban for the prevention of stroke or non-central nervous system (CNS) systemic embolism (SE). Patients must also meet all the eligibility for the study.
Sampling Method: Non-Probability Sample
Enrollment: 493 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Major bleeding events | Up to 12 months

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Up to 12 months
Occurrence of All-cause mortality | Up to 12 months
Occurrence of non-major bleeding events | Up to 12 months
Occurrence of symptomatic thromboembolic events | Up to 12 months
Day(s) of rivaroxaban treatment: start of rivaroxaban therapy and, if applicable, stop of rivaroxaban therapy (in case of treatment discontinuation, switch, or interruption, the reason will be recorded) | Up to 12 months
Changes in creatinine clearance (CrCl) from baseline | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.